CLINICAL TRIAL: NCT05032586
Title: The Effect of Virtual Reality on Pain, Anxiety, and Fear During Burn Dressing in Children: A Randomized Controlled Study
Brief Title: The Effect of Virtual Reality on Pain, Anxiety, and Fear During Burn Dressing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, MERVE KAYA, Ataturk University, Ataturk University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: merve25
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Fear and Anxiety
Keywords: anxiety; burn dressing; child; fear; pain; virtual reality
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: parallel assigment
Masking Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control groups: without wearing virtual reality headsets (No Intervention): Before dressing, the child was given paracetamol, which is routinely used to prevent pain. The child was reminded that they would be with their family during the procedure, and either the mother or father was taken to the dressing room during dressing. After the standard burn dressing was applied to the patient by the healthcare personnel in the burn center treatment room, oxygen saturation and heart rate measurements were made again after the procedure and recorded in the "Application Registration Form." Before and after the procedure, the patients were asked about the pain and anxiety levels felt during dressing and marked on the Wong Baker Scale, State-Trait Anxiety Inventory for Children and Children's Fear Scale.
- experimental groups (Experimental): When the patient adapted to the headset and started to play games, he was taken to the dressing room with the VR headset and the application continued until the process was completed. Before starting the study, a pilot study was conducted to determine the time to wear headsets in ten children. It was observed that the children who were taken to the dressing room without wearing VR headsets refused to wear it. In order to prevent the child from experiencing anxiety in the dressing room, the child was put on VR headset in the patient room and then taken to the dressing room. After the procedure was completed, the VR headset was removed and the patient's oxygen saturation and heart rate were recorded on the "Application Registration Form." The patients were asked regarding the pain and anxiety levels felt during dressing before and after the procedure and marked on the Wong Baker Scale, State-Trait Anxiety Inventory for Children and Children's Fear Scale.
  Interventions: Device: wearing virtual reality headsets

INTERVENTIONS:
Device: wearing virtual reality headsets — When the patient adapted to the headset and started to play games, he was taken to the dressing room with the VR headset and the application continued until the process was completed. Before starting the study, a pilot study was conducted to determine the time to wear headsets in ten children. It was observed that the children who were taken to the dressing room without wearing VR headsets refused to wear it. In order to prevent the child from experiencing anxiety in the dressing room, the child was put on VR headset in the patient room and then taken to the dressing room. After the procedure was completed, the VR headset was removed and the patient's oxygen saturation and heart rate were recorded on the "Application Registration Form." The patients were asked regarding the pain and anxiety levels felt during dressing before and after the procedure and marked on the Wong Baker Scale, State-Trait Anxiety Inventory for Children and Children's Fear Scale.
  Arms: experimental groups

SUMMARY:
This research was conducted to determine the effect of VR on the pain, anxiety, and fear levels experienced by patients during burn dressing. The experimental (VR group) (n=33) and the control group (n=32) were determined using the simple randomization method for the children participating in the study (n=65).

DETAILED DESCRIPTION:
Burn injuries are considered one of the most severe physical and psychosocial traumas a person can face. Burn injuries, especially in the childhood, are an important health problem that causes long-term psychological and physiological consequences and includes rehabilitation processes that continue for years.

During burn treatment, wound debridement, daily dressing change, repair surgeries, and applications during hospitalization cause serious pain, physical stress, and psychological damage to the patient in burn injuries, as in all injuries. Anxiety, loss of control, hopelessness, disruption of body integrity, and pain during burns and procedures during the treatment process are early traumatic features of the burn.

Since pain is not only a sensory experience but also an emotional and cognitive experience, using pharmacological treatment methods alone may not be sufficient. Using nonpharmacological methods in addition to pharmacological methods is recommended in order to control the pain that occurs during wound care and reduce the dose of analgesic administered. The distraction technique is one of the most frequently preferred nonpharmacological methods to reduce pain perception during dressing and control fear and anxiety in children hospitalized in the clinic due to burns. It is a method included in the Nursing Interventions Classification taxonomy.

When the literature was examined, it was observed that there are a limited number of studies examining the effect of VR on pain and anxiety in children during burn dressing. However, there was no study evaluating the fear experienced during burn dressing in children. This study aimed to propagate the use of VR, which is a potentially important technology for nursing care and multidisciplinary healthcare team and has an important place in the treatment of burn patients by reducing the level of pain and anxiety experienced by patients. It is thought that the result of the research will shed light on how to reduce pain, fear, and anxiety experienced during dressing and contribute to the literature as an evidence-based nonpharmacological method.

The research is a randomized controlled experimental study conducted between April 2019 and September 2020. The experimental (VR group) (n=33) and the control group (n=32) were determined using the simple randomization method for the children participating in the study (n=65). The data were collected using the Descriptive Information Form, Wong-Baker FACES Pain Rating Scale, Children's Fear Scale, and State-Trait Anxiety Inventory for Children. In addition, oxygen saturation and heart rate measurements were recorded before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* being in the 7-12 age group,
* not having any dressing in the burn center before
* having a second degree superficial and deep burn
* having burns with a percentage of less than 10%,
* having upper and lower extremity burns
* not having any chronic disease other than burns,
* being willing to participate in the study,
* not having any mental and communication problems and visual impairments

Exclusion Criteria:

* being <7 and >12 years old
* having previous dressing in the burn center,
* having a 1st or 3rd degree burn area,
* having burns on the head, trunk, and genital area,
* having chronic illness other than burns any
* not being willing to participate in the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Descriptive Information Form | up to 1 hour
  The Descriptive Information Form prepared by the researcher consists of 15 questions in total.
Wong-Baker FACES Pain Rating Scale | up to 1 hour
  This scale is used in children aged ≥3 to rate the severity of pain. This numerical rating scale ranges from 0 to 5. Faces show emotions from smiling (0 = very happy/no pain) to crying (5 = hurts worst)
Children's Fear Scale | up to 1 hour
  This scale is a one-item self-report measure for measuring pain-related fear in children. It consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right.
State-Trait Anxiety Inventory for Children (STAI-C) | up to 1 hour
  The scale was transformed into 2 separate scales containing a total of 40 items (20 state and 20 trait anxiety items) as a result of some processes. The scale was seen to be used in all school-age children who can read. The maximum score that can be obtained from the State Anxiety Inventory is 60 and the minimum score is 20

CONTACTS AND LOCATIONS:
Locations (1):
- TURKEY, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No